CLINICAL TRIAL: NCT01992081
Title: A 6-month Multicenter Randomized Trial to Evaluate the Impact of the "PROactive Telecoaching Program" on Physical Activity in Patients With COPD
Brief Title: Study to Evaluate the Impact of the "PROactive Telecoaching Program" on Physical Activity in Patients With COPD.
Acronym: PROactive
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIDD001D2101
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2014-05

CONDITIONS: COPD
Keywords: COPD, Physical Activity, Telecoaching, PROactive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telecoaching (Experimental): Participants will receive daily coaching by an automated telehealth system and coaching by the investigator during study visits, in addition to the usual care.
  Interventions: Device: Automated telehealth system; Other: Usual care
- Control (Other): Participants will receive the usual care but will NOT receive daily coaching by telehealth system.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Automated telehealth system — The automated telehealth system (used within its intended use) comprises of CE marked medical devices and a CE marked step counter (Fitbug®), all being used within their intended use. Coaching by investigators is performed during the study visits and is aimed to enhance physical activity in patients across a spectrum of COPD severity, in addition to the usual care.
  Other Names: telehealth system
  Arms: Telecoaching
Other: Usual care — Participants will receive usual care associated with Chronic Obstructive Pulmonary Disease (COPD)

SUMMARY:
This study will test two instruments to measure physical activity in COPD patients: A questionnaire and two small physical activity monitors .Patients will be randomized to either receive the telecoaching program in addition to usual care or only the usual care. Study will include around 510 patients in 5 countries in Europe.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) has a negative influence on physical activity hence it may be beneficial for patients to increase physical activity levels. This study will test two instruments to measure physical activity: A questionnaire (completed on a personal digital assistant) and a physical activity monitor which patient wear during the day. Patients will be randomized to either receive the Telecoaching program in addition to usual care or only the usual care. The study will involve 4 clinic visits as well as some phone calls over duration of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male and female patients ≥ 40 years of age
* Diagnosis of COPD (GOLD criterion: post bronchodilator FEV1/FVC< 70%)
* Current or ex-smokers with a smoking history equivalent to at least 10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year)
* Patients should have at least 4 days of physical activity data recorded via activity monitor during 7 days prior to visit 101.

Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for inclusion in this study.

* Orthopedic, neurological or other complaints that significantly impair normal biomechanical movement patterns, as judged by the investigator. Specifically if the patients' condition/ co-morbidities are such that physical activity cannot be increased.
* Respiratory diseases other than COPD (e.g. asthma)
* Cognitive reading impairment and/or difficulties to manage electronic devices precluding interaction with the health base and PDA, as judged by the investigator
* Participating in or scheduled to start a rehabilitation program during the study. If the patient wishes to participate in pulmonary rehabilitation for any reason the patient can be enrolled in the study only at the end of rehabilitation.
* Women of child-bearing potential who have the intention to become pregnant during the course of the study and pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive β-hCG laboratory test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The impact of telecoaching program on the physical activity | 6 months
  Impact of telecoaching program on the physical activity of COPD patients will be measured via the use of two PROactive monitors (ActiGraph® and DynaPort®) and a PDA to complete the PROactive questionnaire.
The construct validity of the PROactive instrument. | 6 months
  Construct validity of the PROactive instrument will be measured via the use of two PROactive monitors (ActiGraph® and DynaPort®) and a PDA to complete the PROactive questionnaire.
The responsiveness of the PROactive instrument. | 6 months
  Responsiveness of the PROactive instrument will be measured via the use of two PROactive monitors (ActiGraph® and DynaPort®) and a PDA to complete the PROactive questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Innovative Medicines Initiative, Principal Investigator — PROactive is part of the European Innovative Medicines Initiative (IMI)